CLINICAL TRIAL: NCT01940913
Title: Efficacy and Safety of a Probiotic Product in Children With Antibiotic-associated Gastrointestinal Disorders.
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Probi AB (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Prevention
Other Study IDs: ProAAD
Record Dates: First submitted 2013-09-09; First posted 2013-09-12 (Estimated); Last update posted 2014-05-09 (Estimated); Status verified 2014-05

CONDITIONS: Antibiotic-associated Loose/Watery Stools
MeSH Terms: conditions — Diarrhea | interventions — Probiotics

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor

ARMS (2):
- Probiotics (Active Comparator)
  Interventions: Dietary Supplement: Probiotic capsules
- Placebo (Placebo Comparator)
  Interventions: Dietary Supplement: Placebo capsules

INTERVENTIONS:
Dietary Supplement: Probiotic capsules
  Arms: Probiotics
Dietary Supplement: Placebo capsules
  Arms: Placebo

SUMMARY:
To assess the tolerability and effect of a probiotic product, when co-administered with antibiotics, on the incidence and duration of loose/watery stools following the antibiotic treatment in children.

ELIGIBILITY:
Inclusion criteria

1. Children at the age of 1-11 years that have been ordinated to start antibiotic treatment except for penicillin.
2. Possibility to initiate the probiotic treatment within 24 hours after the first dose of the antibiotic treatment.
3. Children whose parents or legal caregivers have signed the informed consent to participate in the study.

Exclusion criteria

1. Chronic intestinal disease.
2. Current immunodeficiency or immunosuppressive treatment.
3. Chronic or acute diarrhoeal disease.
4. Use of laxatives the week before inclusion in the study.
5. Antibiotic treatment for the last four weeks before inclusion in the study.
6. Known hypersensitivity to any of the ingredients in the probiotic product or the placebo [potato starch, silicon dioxide, capsule (hypromellose, water) ± bacterial culture].
7. Intake of any probiotic products for the last two weeks before inclusion in the study.
8. Patient requiring hospitalisation. Lack of parents´/legal guardians´ informed consent.

Ages: 1 Year to 11 Years | Sex: All
Age Groups: Child
Enrollment: 400 (Estimated)
Dates: Start 2013-10; Primary Completion 2014-04 (Actual); Study Completion 2014-05 (Actual)

PRIMARY OUTCOMES:
Reduction of the incidence of loose/watery stools following antibiotic treatment in children. | 19-24 days

CONTACTS AND LOCATIONS:
Locations (1):
- Multicenter study at 13 health care centers in Warsaw, Warsaw, Poland

REFERENCES:
- [Derived] Olek A, Woynarowski M, Ahren IL, Kierkus J, Socha P, Larsson N, Onning G. Efficacy and Safety of Lactobacillus plantarum DSM 9843 (LP299V) in the Prevention of Antibiotic-Associated Gastrointestinal Symptoms in Children-Randomized, Double-Blind, Placebo-Controlled Study. J Pediatr. 2017 Jul;186:82-86. doi: 10.1016/j.jpeds.2017.03.047. Epub 2017 Apr 21. PMID 28438377